CLINICAL TRIAL: NCT00813904
Title: A Phase 4, Open-Label, Single-Group Immunogenicity and Safety Study of Re-exposure to RECOTHROM� (rThrombin) in Surgical Hemostasis
Brief Title: Immunogenicity and Safety Study of rThrombin in Surgical Hemostasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 499G02
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-11

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — recombinant human thrombin; Thrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rThrombin, 1000 IU/mL (Experimental)
  Interventions: Biological: rThrombin, 1000 IU/mL

INTERVENTIONS:
Biological: rThrombin, 1000 IU/mL — At least 1 application of reconstituted rThrombin, 1000 IU/mL, applied topically directly to the bleeding site, per product labeling.
  Other Names: RECOTHROM

SUMMARY:
The objective of this study is to assess the immunogenicity and safety of recombinant Thrombin (rThrombin) in patients with prior rThrombin exposure.

DETAILED DESCRIPTION:
The safety, immunogenicity, and efficacy of rThrombin have been evaluated in Phase 2 and Phase 3 studies in the following surgical indications: spinal surgery, major hepatic resection, peripheral arterial bypass (PAB) surgery, arteriovenous (AV) graft formation for hemodialysis access, and skin graft surgery following burn injury. Limited data on rThrombin reexposure currently exist. This study will assess the immunogenicity and safety of rThrombin in participants who are undergoing a surgical procedure during which topical rThrombin application is planned and who previously received rThrombin in Phase 3 clinical trials or during prior spine, AV graft formation, or PAB surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in a ZymoGenetics-sponsored Phase 3 study and the recipient of treatment with rThrombin in that study or the recipient of commercially-available rThrombin in a prior spine, arteriovenous graft formation, or peripheral artery bypass surgical procedure
* Age of 18 years or older at time of consent
* Bleeding indicating treatment with rThrombin during the course of the surgical procedure
* Signed informed consent document approved by an institutional review board or independent ethics committee

Exclusion Criteria:

* Currently undergoing a procedure requiring cardiopulmonary bypass or involving the aortic arch
* Known hypersensitivity to rThrombin product or any of its components
* Currently undergoing a surgical procedure where the use of other thrombin-containing hemostatic agents is planned
* Medical, social, or psychosocial factors that, in the opinion of the investigator, could affect the participant's safety or compliance with study procedures
* Treatment with any experimental agent within 30 days of study enrollment or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Principal Investigator — Lotus Clinical Research
Locations (1):
- Tuscon Orthopaedic Institute, Tuscon, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 31 participants enrolled, all received treatment with recombinant thrombin (rThrombin).
Groups:
- rThrombin, 1000 IU/mL: At least 1 application of reconstituted rThrombin, 1000 IU/mL, applied topically directly to the bleeding site.
Period: Overall Study
Arm/Group | rThrombin, 1000 IU/mL
Started | 31
Completed | 30
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 31
Age, Customized [Mean (Standard Deviation); unit: Years] | 59.5 (12.3)
Age, Customized [Median (Full Range); unit: Years]
  Median | 61.0 [22.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Type of surgery [Number; unit: Participants]
  Arterial reconstruction/peripheral arterial bypass | 4
  Arteriovenous vascular access procedure | 3
  Other | 1
  Spinal | 23

OUTCOME MEASURES:

1. Primary Outcome: Number or Participants With Antirecombinant Thrombin (rThrombin) Product Antibody at Baseline and Day 29
Description: Immunogenicity of rThrombin product was evaluated using an enzyme-linked immunosorbent assay for detection of antirThrombin product antibody and a neutralizing antibody assay to characterize the potential of antibodies to rThrombin product to neutralize the activity of human plasma-derived thrombin.
Time Frame: At baseline and Day 29
Population: Participants who received treatment with rThrombin and had data available from both baseline and Day 29 antibody assessments.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 30
Participants
  Baseline | 0
  Day 29 | 0

2. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, Adverse Events (AEs), Treatment-related Adverse Events, and AEs Leading to Discontinuation
Description: An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. Treatment-related=possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: Baseline through Day 29, continuously
Population: All participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 31
Participants
  Death | 1
  SAEs | 6
  Treatment-related SAEs | 0
  AEs | 29
  Treatment-related AEs | 0
  AEs leading to discontinuation | 0

3. Secondary Outcome: Number of Participants With AEs by Maximum Severity
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. AE severity was assessed using Common Terminology Criteria for Adverse Events, Version 13.0: Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening; Grade 5=fatal.
Time Frame: Baseline to Day 29, continuously
Population: All participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 31
Participants
  Mild | 1
  Moderate | 18
  Severe | 9
  Life-threatening | 0
  Fatal | 1

ADVERSE EVENTS:
Arm/Group | TOTAL
Serious Adverse Events (participants affected / at risk) | 6/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TOTAL (N=31)
CHEST PAIN (General disorders) | 1
OSTEOMYELITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 1
SYNCOPE (Nervous system disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1
HYPOTENSION (Vascular disorders) | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TOTAL (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 2
TACHYCARDIA (Cardiac disorders) | 6
CONSTIPATION (Gastrointestinal disorders) | 8
NAUSEA (Gastrointestinal disorders) | 8
VOMITING (Gastrointestinal disorders) | 2
PYREXIA (General disorders) | 3
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 6
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 5
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 3
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 23
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
HYPOAESTHESIA (Nervous system disorders) | 2
RADICULOPATHY (Nervous system disorders) | 2
INSOMNIA (Psychiatric disorders) | 4
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 4
HYPERTENSION (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZymoGenetics (ZG) agreements vary by trial, but each states that presentation/publication (p/p) cannot disclose Confidential Information (CI), excluding trial results; p/p may not begin until the earlier of 18 months after study end, ZG/lead investigator publishes, or ZG notification that multicenter publication is not planned; ZG has specified time for draft review before submission/presentation and may delay or modify content, require CI removal, and delay p/p for patent application filing.